CLINICAL TRIAL: NCT04496739
Title: Cluster Randomized Controlled Trial of Patient and Provider Decision Support to Increase Chemoprevention Informed Choice Among Women With Atypical Hyperplasia or Lobular Carcinoma In Situ - Making Informed Choices on Incorporating Chemoprevention Into Care (MiChoice)
Brief Title: Making Informed Choices on Incorporating Chemoprevention Into Care (MiCHOICE)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S1904; NCI-2019-08755 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1904 (Other: SWOG); SWOG-S1904 (Other: DCP); S1904 (Other: CTEP); R01CA226060 (NIH); UG1CA189974 (NIH)
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Atypical Hyperplasia of the Breast; Lobular Breast Carcinoma In Situ; Pleomorphic Lobular Breast Carcinoma In Situ
MeSH Terms: conditions — Breast Carcinoma In Situ | interventions — Decision Support Techniques; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (educational materials) (Active Comparator): Patients receive standard educational materials about breast cancer risk and chemoprevention in RealRisks via the patient portal or website.
  Interventions: Behavioral: Cancer Educational Materials; Other: Questionnaire Administration
- Group II (educational materials, decision support, interview) (Experimental): Patients receive standard educational materials about breast cancer risk and chemoprevention in RealRisks via the patient portal or website. Patients receive patient-centered decision support within the patient portal via an action plan summarizing their breast cancer risk profile, their risks and benefits of SERMs and AIs, and personal preferences for chemoprevention. Health care providers receive decision support and action plans based on their patients' interactions with RealRisks via the BNAV provider-centered support tool within the EHR. A sample of patients participate in an audio-recorded interview via telephone or video conference over 45-60 minutes at 12 months after registration. A sample of health care providers participate in 3 audio-recorded interviews via telephone or video conference over 45-60 minutes each at baseline, within 12-36 months after study activation, and within 12 months after study closure to accrual.
  Interventions: Behavioral: Cancer Educational Materials; Other: Decision Aid; Other: Interview; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Cancer Educational Materials — Receive educational materials about breast cancer risk and chemoprevention via RealRisk
Other: Decision Aid — Given patient-centered decision support via an action plan
  Arms: Group II (educational materials, decision support, interview)
Other: Decision Aid — Given decision support and action plans based on patient's interactions with RealRisks via the BNAV support tool
  Arms: Group II (educational materials, decision support, interview)
Other: Interview — Participate in audio-recorded interview via telephone or video conference
  Arms: Group II (educational materials, decision support, interview)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies the implementation of web-based decision support tools for patients with atypical hyperplasia or lobular carcinoma in situ and healthcare providers. Decision support tools are designed to improve informed choice about breast cancer chemoprevention. Recognizing barriers and facilitators that can influence the adoption of decision support tools at recruitment centers may help researchers learn how to best implement them into clinical practice.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the frequency of chemoprevention informed choice at 6 months after registration among women with atypical hyperplasia (AH) or lobular carcinoma in situ (LCIS) between the intervention (RealRisks decision aid/breast cancer risk navigation [BNAV] + standard educational materials) and control (standard educational materials alone) arms.

SECONDARY OBJECTIVES:

I. To assess patient chemoprevention knowledge, chemoprevention intention/decision, perceived breast cancer risk and worry, accuracy of breast cancer risk perception, decision conflict and decision regret at baseline, 6 months, and 12 months in the intervention and control arms.

II. To compare patient chemoprevention usage, adherence, and reasons for discontinuation of a selective estrogen receptor modulator (SERM) or aromatase inhibitor (AI) annually for up to 5 years between the intervention and control arms.

III. To assess shared decision-making about chemoprevention among patients and healthcare providers after their 6-month clinic visit in the intervention and control arms.

IMPLEMENTATION OBJECTIVE:

I. To assess the implementation of the decision support tools, RealRisks and BNAV, into clinic workflow, and to better understand barriers and facilitators to chemoprevention usage by conducting telephone/video-conference interviews of healthcare providers and high-risk women with AH or LCIS assigned to the active intervention.

OUTLINE: Recruitment centers are randomized to 1 of 2 groups.

GROUP I (CONTROL): Patients receive standard educational materials about breast cancer risk and chemoprevention in RealRisks via the patient portal or website.

GROUP II (INTERVENTION): Patients receive standard educational materials about breast cancer risk and chemoprevention in RealRisks via the patient portal or website. Patients receive patient-centered decision support within the patient portal via an action plan summarizing their breast cancer risk profile, their risks and benefits of SERMs and AIs, and personal preferences for chemoprevention. Health care providers receive decision support and action plans based on their patients' interactions with RealRisks via the BNAV provider-centered support tool within the electronic health record (EHR). A sample of patients participate in an audio-recorded interview via telephone or video conference over 45-60 minutes at 12 months after registration. A sample of health care providers participate in 3 audio-recorded interviews via telephone or video conference over 45-60 minutes each at baseline, within 12-36 months after study activation, and within 12 months after study closure to accrual.

After completion of study, patients are followed up at 6, 12, 24, 36, 48, and 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically-confirmed atypical hyperplasia (AH) or lobular carcinoma in situ (LCIS) documented by breast pathology report at any time in the past. Patients with borderline breast lesions and pleomorphic LCIS are also eligible
* Patients must be women at least 35 and no more than 74 years of age at registration, since the Breast Cancer Surveillance Consortium (BCSC) risk calculator is valid only for this age range
* Both pre/perimenopausal and postmenopausal women are eligible
* Patients must be able to read and write in English or Spanish since study questionnaires and educational materials are only available in English and Spanish
* Baseline questionnaires must be completed prior to patient registration
* The S1904 Patient Contact form must be completed prior to patient registration
* Patients must be able to access the internet and receive email or text messages. This is required to access study materials and receive email/text message reminders from the S1904 Study Team at Columbia University Irving Medical Center (CUIMC). The patient decision aid, RealRisks, is accessible via smartphones, tablets, or personal computers. If patients do not own these devices, local study personnel will provide resources for patients to access RealRisks via computer kiosks or tablets in clinic waiting rooms or public locations, such as community centers or public libraries
* Patients and healthcare providers must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* IMPLEMENTATION: Providers who enrolled in S1904 at Group 2 (intervention) recruitment center and consented to future contact are eligible to participate in the interviews
* IMPLEMENTATION EVALUATION: Patients who registered to S1904 at a Group 2 (Intervention) Recruitment Center and consented to be contacted for future research are eligible to participate in the interviews
* Recruitment Centers must be National Clinical Trials Network (NCTN), National Cancer Institute Community Oncology Research Program (NCORP) or Minority Underserved (MU)-NCORP institutions
* Recruitment Centers must have an active EHR and patient portal used in the outpatient clinics which is common and accessible across all sites belonging to the Recruitment Center
* Recruitment Centers must be willing to allow the S1904 study team access to the site's application program interface (API) for integration of the study materials (standard educational materials and decision support tools) into the EHR and patient portal. (NOTE: Both Group 1 (control) and Group 2 (intervention) recruitment centers may access the standard educational materials via the patient portal or uniform resource locator (URL)/website)
* Recruitment centers must see at least 50 AH and/or LCIS patients per year
* Recruitment centers must identify a lead principal investigator (PI) to facilitate recruitment and retention of patients and healthcare providers and to participate in quarterly stakeholder meetings/conference calls
* Recruitment centers must be willing to register at about 16 patients and 5 healthcare providers to the study
* Recruitment Centers must be willing to submit monthly screening logs to CUIMC
* Providers must regularly see patients with AH or LCIS at an approved recruitment center
* Providers must be willing to provide informed consent and complete an online baseline questionnaire
* Providers who will register patients must be registered members of a Cooperative Group
* Providers who register patients to S1904 must be willing to see those same patients for their 6-month study visits, as the provider intervention tools require that the "treating investigator" as designated in OPEN and the provider at the 6-month study visit be the same

Exclusion Criteria:

* Patients must not have a history of invasive breast cancer or ductal carcinoma in situ
* Patients must not have prior or current use of selective estrogen receptor modulators (SERMs) or aromatase inhibitors (AIs)

  * NOTE: The following are approved SERMS and AIs, however, the study is not limited to these.

    * SERMs: tamoxifen, raloxifene
    * AIs: anastrozole, exemestane, letrozole
* Patients must not be currently taking hormone replacement therapy
* Patients must not have a history of bilateral mastectomies or breast implants since the risk calculator is not applicable to these women
* Patients must not be pregnant or lactating
* Premenopausal patients must not have a history of thromboembolism, since it is a contraindication to tamoxifen. Tamoxifen is the only Food and Drug Administration (FDA)-approved drug for breast cancer chemoprevention among high-risk premenopausal women, whereas postmenopausal women are eligible for both SERMs and AIs

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Chemoprevention informed choice | At 6 months
  Will be provided by chemoprevention knowledge scale, a 1-item attitudes scale, and chemoprevention decision and measure at 6 and 12 months on the S1904 Follow-Up Choice form. All enrolled patients who provide outcomes data at the 6-month timepoint will be included in the primary analysis under the intention-to-treat principle. The primary analysis of the intervention effect on informed choice at 6 months will be based on a logistic regression model using a generalized estimating equation approach to account for clustering. Additional supportive analyses will adjust for both patient and clinic level factors. If there are substantial missing data for the components of the primary endpoint, a sensitivity analysis will be conducted imputing a response of no informed decision making for those women with missing information.

SECONDARY OUTCOMES:
Perceived breast cancer risk | Up to 12 months
  Will be assessed by absolute estimate ("How do you rate your chance of developing breast cancer?"), comparative risk ("Overall, how do you think your chance of developing breast cancer compares to the average woman your age?"), and numeric risk ("Please place an X on the line below at the point showing what you think your chance is of developing breast cancer in the next five years"). All are assessed on a scale of 0% to 100%, with 0% as "no chance of breast cancer" and 100% as "definitely will get breast cancer."
Actual breast cancer risk score | Up to 12 months
  A numeric score between the values of 0% and 100%, as determined by the Breast Cancer Surveillance Consortium (BCSC) risk models. The 5-year and 10-year risk estimates are used. The items needed for the BCSC risk models are obtained at baseline from the S1904 Onstudy.
Accuracy of risk perception | Up to 12 months
  Will be defined as the difference between numeric perceived breast cancer 10-year risk estimate (subjective) and actual 10-year breast cancer risk score, according to the BCSC risk model (objective). Categorized as: accurate if the difference between subjective and objective risk estimates are =< 10% in either direction; underestimate if > 10% below objective risk; and overestimate if > 10% above objective risk.
Breast cancer worry | Up to 12 months
  Will be measured by two Likert-style items, with responses ranging from "Not at all" (1) to "All of the time" (7). Items are reported and scored separately. Breast cancer worry is assessed on the S1904 Breast Cancer Risk Questionnaire.
Decision conflict | Up to 12 months
  Will be assessed on the S1904 Breast Cancer Risk Questionnaire. Will be measured by a validated 10-item scale with 3 response categories (Yes/Unsure/No) to assess the level of conflict women feel about their decisions regarding chemoprevention. Scores range from 0 (no decisional conflict) to 100 (extremely high decisional conflict) and will be scored according to the User Manual - Decisional Conflict Scale.
Decision regret | Up to 12 months
  Will be assessed on the S1904 Decision Questionnaire. Will be measured by a validated 5-item scale composed of 5-point Likert-style items. Scores that range from 0 (no regret) to 100 (high regret). It is scored according to the User Manual - Decision Regret Scale.
Chemoprevention usage | Up to 5 years
  Will be assessed on the S1904 Follow-Up form and the S1904 Breast Cancer Risk-Reducing Pill Usage form. Among patients who do not have a diagnosis of invasive breast cancer or ductal carcinoma in situ, it will be defined as reporting having started taking or currently taking a selective estrogen receptor modulators (SERM) or aromatase inhibitor (AI) for primary prevention, as assessed by self-report, and taking at least one dose of a SERM or AI for primary prevention, as assessed by the site based on the electronic health record log. Both measures will be reported. Reasons for never starting chemoprevention will be recorded.
Chemoprevention adherence | Up to 5 years
  Will be assessed using a 3-item scale for patients currently taking a SERM or AI. Responses are given values 1 through 5, with the response corresponding to perfect adherence assigned 1. The three scores are averaged if at least 2 of the 3 items have responses. Non-adherence is defined as an average score of greater than 1. Will be assessed on the S1904 Breast Cancer Risk-Reducing Pill Usage form.
Reasons for chemoprevention discontinuation | Up to 5 years
  For patients who report discontinuing a SERM or AI, reasons for discontinuing chemoprevention are reported on the S1904 Breast Cancer Risk-Reducing Pill Usage form.
Shared decision-making | Up to 6 months
  Will be assessed by a validated 9-item scale with Likert-style responses to assess shared decision-making about chemoprevention. Scores range from 0 to 100. Provider and patient measures are evaluated separately and scored according to their respective validation papers. Will be assessed on the S1904 Patient Shared Decision-Making Questionnaire and on the S1904 Provider Shared Decision-Making Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine D Crew, Principal Investigator — SWOG Cancer Research Network
Locations (97):
- United States (96):
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - UC Irvine Health Cancer Center-Newport, Costa Mesa, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Miami Cancer Institute, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Miami Cancer Institute at Plantation, Plantation, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Diagnostic Radiology Services LLC, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Straub Medical Center - Kahului Clinic, Kahului, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Loyola Center for Health at Burr Ridge, Burr Ridge, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - IU Health West Hospital, Avon, Indiana
  - IU Health North Hospital, Carmel, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Beverly Hospital, Beverly, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Winchester Hospital, Winchester, Massachusetts
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, East White Plains, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Good Samaritan Hospital, Corvallis, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Holy Redeemer Hospital and Medical Center, Meadowbrook, Pennsylvania
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Baptist Memorial Hospital for Women, Memphis, Tennessee
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Peninsula Cancer Institute-Newport News, Newport News, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Shenandoah Oncology PC, Winchester, Virginia
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
- FHP Health Center-Guam, Tamuning, Guam

REFERENCES:
- [Derived] Michel AM, Yi H, Amenta J, Collins N, Vaynrub A, Umakanth S, Anderson G, Arnold K, Law C, Pruthi S, Sandoval-Leon A, Shirley R, Perdekamp MG, Colonna S, Krisher S, King T, Yee LD, Ballinger TJ, Braun-Inglis C, Mangino DA, Wisinski K, DeYoung CA, Ross M, Floyd J, Kaster A, VanderWalde L, Saphner TJ, Zarwan C, Lo S, Graham C, Conlin A, Yost K, Agnese D, Jernigan C, Hershman DL, Neuhouser ML, Arun B, Crew KD, Kukafka R. Use of web-based decision support to improve informed choice for chemoprevention: a qualitative analysis of pre-implementation interviews (SWOG S1904). BMC Med Inform Decis Mak. 2024 Sep 27;24(1):272. doi: 10.1186/s12911-024-02691-0. PMID 39334347
- [Derived] Crew KD, Anderson GL, Arnold KB, Stieb AP, Amenta JN, Collins N, Law CW, Pruthi S, Sandoval-Leon A, Bertoni D, Grosse Perdekamp MT, Colonna S, Krisher S, King T, Yee LD, Ballinger TJ, Braun-Inglis C, Mangino D, Wisinski KB, DeYoung CA, Ross M, Floyd J, Kaster A, Vander Walde L, Saphner T, Zarwan C, Lo S, Graham C, Conlin A, Yost K, Agnese D, Jernigan C, Hershman DL, Neuhouser ML, Arun B, Kukafka R. Making Informed Choices On Incorporating Chemoprevention into carE (MiCHOICE, SWOG 1904): Design and methods of a cluster randomized controlled trial. Contemp Clin Trials. 2024 Jul;142:107564. doi: 10.1016/j.cct.2024.107564. Epub 2024 May 3. PMID 38704119
- [Derived] McGuinness JE, Bhatkhande G, Amenta J, Silverman T, Mata J, Guzman A, He T, Dimond J, Jones T, Kukafka R, Crew KD. Strategies to Identify and Recruit Women at High Risk for Breast Cancer to a Randomized Controlled Trial of Web-based Decision Support Tools. Cancer Prev Res (Phila). 2022 Jun 2;15(6):399-406. doi: 10.1158/1940-6207.CAPR-21-0593. PMID 35412592